CLINICAL TRIAL: NCT00260858
Title: Measuring the Glycaemic Index of Foods: Interlaboratory Study #2
Brief Title: GI Interlab 2 Study: Measuring the Glycaemic Index (GI) of Foods
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Glycaemic Index Testing, Inc. (Industry)
Collaborators: Sydney University Glycaemic Index Research Services (Unknown); ILSI Europe (Unknown)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: GIL5047
Record Dates: First submitted 2005-11-30; First posted 2005-12-02 (Estimated); Last update posted 2006-06-09 (Estimated); Status verified 2006-06

CONDITIONS: Healthy
Keywords: Glycemic index; Nutrition; Carbohydrates; Glycemic responses; Methodology; Healthy human subjects
MeSH Terms: interventions — Glucose

INTERVENTIONS:
Drug: Test Meal: Reference food (glucose or white bread)
Drug: Test Meal: Pirate's Booty
Drug: Test Meal: Ceaprove wafer
Drug: Test Meal: Stretch Island Strawberry Fruit Leather

SUMMARY:
The purpose of this study is to assess the extent of and sources of variation in the glycaemic index values of foods measured by different laboratories around the world.

DETAILED DESCRIPTION:
The glycaemic index values of 3 different foods provided from a central location will be determined in each of 20-30 centers around the world. A standard protocol will be followed, but this protocol leaves room for variation in certain details, such as whether subjects are allowed to have coffee or tea with the test meals or only water, or the method of analyzing blood glucose. Methodologic details, subject demographic information (height, weight, age, and ethnicity), results of local calculations and raw data will be sent to a central location.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male or female subjects

Exclusion Criteria:

* Diabetes
* Pregnancy or lactation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 280
Dates: Start 2005-11; Study Completion 2006-04

PRIMARY OUTCOMES:
glycaemic index

SECONDARY OUTCOMES:
within-individual variation of glycaemic responses
glycaemic responses assessed as incremental area under the curve

CONTACTS AND LOCATIONS:
Overall Officials: Thomas MS Wolever, MD, PhD, Principal Investigator — University of Toronto; Janette C Brand-Miller, PhD, Principal Investigator — University of Sydney
Locations (28):
- United States (3):
  - Abernethy Research, Gainsville, Florida
  - University of Buffalo, Buffalo, New York
  - Ohio State University, Columbus, Ohio
- Australia (2):
  - University of Sydney, Sydney, New South Wales
  - International Diabetes Institute, Melbourne, Victoria
- Glycemic Index Laboratories, Inc., Toronto, Ontario, Canada
- Institute of Nutrition and Food Safety, Chinese Centre for Disease Control and Prevention, Beijing, Beijing Municipality, China
- The Royal Veterinary & Agricultural University, Copenhagen, Denmark
- Finland (2):
  - National Public Health Institute, Helsinki, Helsinki
  - Foodfiles Oy, Kuopio, Kuopio
- Biofortis, Nantes, Nantes, France
- German Institute of Human Nutrition, Potsdam-Rehbrucke, Nuthetal, Germany
- Italy (2):
  - University of Milan, Milan, Milan
  - University of Parma, Parma, Parma
- University Sains Malaysia, Kota Bharu, Kelantan, Malaysia
- Nutriscience, BV, Maastricht, Maastricht, Netherlands
- University of Otago, Dunedin, Otago, New Zealand
- University of the Philippines, Diliman, Philippines
- South Africa (2):
  - GI Foundation of South Africa, Mbombela, Mpumalanga
  - Potchefstroom University, Potchefstroom, Potchesfstroom
- Sweden (2):
  - Gotheburg University, Gothenburg, Gotheburg
  - Lund University, Lund, Lund
- University of the West Indies, Champs Fleurs, Trinidad, Trinidad and Tobago
- United Kingdom (5):
  - Reading Scientific Services, Ltd., Reading, Berkshire
  - Hammersmith Hospital, London, London
  - Oxford Brookes University, Oxford, Oxfordshire
  - University of Surrey, Guildford, Surrey
  - Leatherhead Food International, Leatherhead, Surrey

REFERENCES:
- [Derived] Wolever TM, Brand-Miller JC, Abernethy J, Astrup A, Atkinson F, Axelsen M, Bjorck I, Brighenti F, Brown R, Brynes A, Casiraghi MC, Cazaubiel M, Dahlqvist L, Delport E, Denyer GS, Erba D, Frost G, Granfeldt Y, Hampton S, Hart VA, Hatonen KA, Henry CJ, Hertzler S, Hull S, Jerling J, Johnston KL, Lightowler H, Mann N, Morgan L, Panlasigui LN, Pelkman C, Perry T, Pfeiffer AF, Pieters M, Ramdath DD, Ramsingh RT, Robert SD, Robinson C, Sarkkinen E, Scazzina F, Sison DC, Sloth B, Staniforth J, Tapola N, Valsta LM, Verkooijen I, Weickert MO, Weseler AR, Wilkie P, Zhang J. Measuring the glycemic index of foods: interlaboratory study. Am J Clin Nutr. 2008 Jan;87(1):247S-257S. doi: 10.1093/ajcn/87.1.247S. PMID 18175765